CLINICAL TRIAL: NCT00496938
Title: A Clinical Evaluation of the XIENCE Everolimus Eluting Coronary Stent System in the Treatment of Women With de Novo Coronary Artery Lesions
Brief Title: XIENCE V: SPIRIT WOMEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-377
Record Dates: First submitted 2007-07-03; First posted 2007-07-06 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Stenosis; Coronary Arteriosclerosis; Coronary Artery Disease; Coronary Artery Restenosis; Total Coronary Occlusion; Stent Thrombosis; Vascular Disease; Myocardial Ischemia
Keywords: Stents; Angioplasty; Total coronary occlusions; Coronary restenosis; Stent thrombosis; Everolimus
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Observational cohort using an all-comers design
  Interventions: Device: XIENCE V®/ XIENCE PRIME™

INTERVENTIONS:
Device: XIENCE V®/ XIENCE PRIME™ — Coronary artery placement of a XIENCE V®/ XIENCE PRIME™ Everolimus Eluting Stent System

SUMMARY:
The purpose of this Clinical Evaluation is the continued assessment of the XIENCE Everolimus Eluting Coronary Stent System (XIENCE V® and XIENCE PRIME™ EECSS) with the primary focus on clinical outcomes in the treatment of female patients with de novo coronary artery lesions, and the characterization of the female population undergoing stent implantation with a XIENCE stent.

DETAILED DESCRIPTION:
SPIRIT Women Single-Arm Study: A prospective, open label, single arm, multi-center study evaluating performance of the XIENCE V® and XIENCE PRIME™ EECSS in the treatment of female patients with coronary artery lesions, per its Instructions for Use (IFU).

The long term safety and efficacy of the XIENCE V EECSS have been demonstrated in the SPIRIT FIRST trial up to 5 years, the SPIRIT II trial up to 4 years, and in the SPIRIT III Randomized Control Trial (RCT) up to 3 years. In addition, these pre-approval studies have shown low rates of Target Vessel Failure and Major Adverse Cardiac Events (MACE) that were observed to plateau or gradually decline after about 1 year and were consistently lower than the comparator arm of each study. This benefit in MACE is sustained for up to 5 years and is also independent of the first year results.

The post approval SPIRIT V study demonstrated that the use of the XIENCE EECSS in complex lesions in a real-world population resulted in 1 year MACE, Stent Thrombosis and Target Lesion Revascularization rates that are comparable to those of the previously mentioned pre-approval studies which included patients with more restricted inclusion / exclusion criteria.

Therefore, based on existing data from these trials, Abbott Vascular has decided to discontinue further follow up in the SPIRIT Women study after 2 years.

ELIGIBILITY:
General Inclusion Criteria:

* Patient must be female.
* Patient must be at least 18 years of age.
* Patient is able to verbally confirm understanding of risks, benefits and treatment alternatives and she or her legally authorized representative provides written informed consent prior to any study related procedure, as approved by the appropriate Medical Ethics Committee of the respective clinical site.
* Patient must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia).
* Patient must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
* Patient must agree to undergo all CIP-required follow-up examinations.
* Patients of childbearing potential must have had a negative pregnancy test within 7 days before treatment, and must not be nursing at the time of treatment.

Angiographic Inclusion Criteria:

* Patients' artery morphology and disease is suitable to be optimally treated with a maximum of 4 planned study stents.
* Target lesions must be de novo lesions (no prior stent implant, no prior brachytherapy).
* Target vessel reference diameter must be between 2.5 mm and 4.0 mm by visual estimate. The diameter range will be expanded to 2.25 mm when the 2.25 mm stent is available.
* Target lesion greater than or equal to 28 mm in length by visual estimate.

General Exclusion Criteria:

* Patient has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the clinical investigation plan, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
* Patient has a known hypersensitivity or contraindication to aspirin, either heparin or bivalirudin, both clopidogrel and ticlopidine, everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
* Participation in another device or drug study or has completed the follow-up phase of another study within the last 30 days.
* Patient who is judged to have a lesion that prevents complete inflation of an angioplasty balloon.
* Patient has had a previous stent implant, either Bare Metal Stent (BMS) or Drug Eluting Stent (DES) within the target vessel(s)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Adjudicated Composite rate of all Death, all Myocardial Infarction (MI) and Target Vessel Revascularization (TVR) | at 1 year

SECONDARY OUTCOMES:
Acute Success (Clinical Device Success and Clinical Procedure Success) | Acute
Adjudicated Stent Thrombosis (Definite, Probable, Possible) | at 30 days
Adjudicated revascularization (TLR/TVR/all revascularizations) | at 30 days
Adjudicated Composite rate of Cardiac Death, MI attributed to the target vessel and CI-TLR. | at 30 days
Adjudicated Composite rate of all Death, all MI and Target Vessel Revascularization (TVR). | at 30 days
Adjudicated Composite rate of all Death, all MI and all Revascularization (TLR/TVR/non TVR. | at 30 days
Adjudicated Cardiac Death, Non-Cardiovascular Death, Vascular Death, Q-wave MI and Non Q-wave MI (Peri-Procedural, Unrelated to PCI). | at 30 days
Adjudicated Stent Thrombosis (Definite, Probable, Possible) | at 240 Days
Adjudicated Stent Thrombosis (Definite, Probable, Possible) | at 1 Year
Adjudicated Stent Thrombosis (Definite, Probable, Possible) | at 2 Years
Adjudicated revascularization (TLR/TVR/all revascularizations) | at 240 Days
Adjudicated revascularization (TLR/TVR/all revascularizations) | at 1 year
Adjudicated revascularization (TLR/TVR/all revascularizations) | at 2 years
Adjudicated Composite rate of Cardiac Death, MI attributed to the target vessel and CI-TLR. | at 240 Days
Adjudicated Composite rate of Cardiac Death, MI attributed to the target vessel and CI-TLR. | at 1 Year
Adjudicated Composite rate of Cardiac Death, MI attributed to the target vessel and CI-TLR. | at 2 Years
Adjudicated Composite rate of all Death, all MI and Target Vessel Revascularization (TVR). | at 240 Days
Adjudicated Composite rate of all Death, all MI and Target Vessel Revascularization (TVR). | at 1 Year
Adjudicated Composite rate of all Death, all MI and Target Vessel Revascularization (TVR). | at 2 Years
Adjudicated Composite rate of all Death, all MI and all Revascularization (TLR/TVR/non TVR. | at 240 Days
Adjudicated Composite rate of all Death, all MI and all Revascularization (TLR/TVR/non TVR. | at 1 Year
Adjudicated Composite rate of all Death, all MI and all Revascularization (TLR/TVR/non TVR. | at 2 years
Adjudicated Cardiac Death, Non-Cardiovascular Death, Vascular Death, Q-wave MI and Non Q-wave MI (Peri-Procedural, Unrelated to PCI). | at 240 Days
Adjudicated Cardiac Death, Non-Cardiovascular Death, Vascular Death, Q-wave MI and Non Q-wave MI (Peri-Procedural, Unrelated to PCI). | at 1 year
Adjudicated Cardiac Death, Non-Cardiovascular Death, Vascular Death, Q-wave MI and Non Q-wave MI (Peri-Procedural, Unrelated to PCI). | at 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Morice, Principal Investigator — Institut Cardiovasculaire Paris Sud (ICPS), Paris, France; Stephan Windecker, Principal Investigator — University Hospital Bern, Bern, Switzerland
Locations (95):
- Argentina (2):
  - Hosital Italiano de Buenos Aires - Cardiologia, Buenos Aires, Buenos Aires
  - Instituto Cardiovascular de Buenos Aires-ICBA, Buenos Aires
- Australia (2):
  - The Northern Hospital, Epping
  - Liverpool Hospital, New South Wales
- Austria (3):
  - Landesklinikum St. Pölten, Sankt Pölten
  - Allgemeines Krankenhaus der Stadt Wien - Univ.Klinik f. Innere Medizin II, Vienna
  - Klinikum Kreuzschwestern Wels GmbH, Wels
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - CHU Charleroi, Charleroi
  - Heilig Hart Ziekenhuis Roeselare, Roeselare
- Brazil (4):
  - Hospital Madre Teresa, Belo Horizonte
  - Hospital Moinhos de Ventos-Centro de Cardiologia, Porto Alegre
  - Instituto de Cardiologia Dante Pazzanese Unidadae II Recepcao de Angioplastia, São Paulo
  - INCOR/SP Instituto do Coração - Hospital das Clinicas - FMUSP, São Paulo
- China (9):
  - Queen Elizabeth Hospital, Hong Kong, Hong Kong
  - Queen Mary Hospital, Hong Kong, Hong Kong
  - Tuen Mun Hospital, Hong Kong, Hong Kong
  - Fu Wai Hospital, Beijing
  - China People Liberation Army (PLA) General Hospital, Beijing
  - Guangzhou Army General Hospital, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - United Christian Hospital, Hong Kong
  - Shanghai Renji Hospital (East), Shanghai
- Rigshospitalet, Copenhagen, Denmark
- France (8):
  - Hôpital Henri Duffaut, Avignon
  - Clinique Saint Augustin, Bordeaux
  - Hôpital de la Cavale Blanche, Brest
  - Hôpital du Bocage - CHU, Dijon
  - Institut Hospitalier Jacques Cartier Service d'Angiographie, Inst Cardiovasculaire Paris-Sud, Massy
  - Hôpital Arnaud de Villeneuve - CHU, Montpellier
  - Centre Cardio-Pneumologique - Hôpital Pontchaillou - CHU, Rennes
  - Hôpital Charles Nicolle, Rouen
- Germany (11):
  - Kardiologische Klinik Herz- und Diabeteszentrum, Bad Oeynhausen
  - Segebergerkliniken, Bad Segeberg
  - Klinikum Coburg GmbH, Coburg
  - Amper Kliniken-Kreisklinik, Dachau
  - Technische Universität Dresden, Medizinische Klinik II - Kardiologie, Dresden
  - Universitäres Herzzentrum, Medizinische Klinik III, Hamburg
  - Medizinische Hochschule Hannover Abteilung Kardiologie Und Angiologie, Hanover
  - Klinikum Ludwigshafen, Ludwigshafen
  - Klinikum der Johannes Gutenberg-Universität II. Medizinische Klinik und Poliklinik, Mainz
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Kliniken Villingen, Villingen-Schwenningen
- Greece (2):
  - Onassis Cardiac Surgery Hospital, Athens
  - Cardiology Clinic of Papageorgiou Hospital, Thessaloniki
- Hungary (2):
  - Semmelweis University, Department of Cardiovascular Surgery, Budapest
  - University of Pécs/Medical School/Heart Institute, Pécs
- India (5):
  - Apollo Hospital, Hyderabaad, Andhar Pradesh
  - CARE Hospital, Hyderabaad, Andhra Pradesh
  - Sanjay Gandhi Postgraduate Institute of Medical Sciences, Lucknow
  - Max Devki Devi Heart & Vascular Insititute, Department of Cardiology, New Delhi
  - Escorts Heart Institute & Research Centre, New Delhi
- Wolfson Medical Center, Holon, Israel
- Italy (12):
  - Ospedale A. Manzoni, Lecco
  - Centro Cardiologico Monzino, Milan
  - Clinico S.Ambrogio, GRUPPO OSPEDALIERO SAN DONATO, Milan
  - Azienda Policlinico di Modena U.O. Cardiologia, Ospedale di Modena, Modena
  - Hesperia Hospital, Modena
  - L'Azienda di Rilievo Nazionale di Alta Specializzazione (A.R.N.A.S.) Civico e Benfratelli, Palermo
  - A.O Di Perugia, Ospedale Silvestrini, Perugia
  - Ospedale Cisanello, Pisa
  - Azienda Ospedaliera Santa Maria Nuova, Reggio Emilia
  - A.O. Universitaria Tor Vergata, Cardiologia, Rome
  - Istituto Clinico Humanitas, Rozzano
  - Instituto Policlinico S. Donato, San Donato
- Latvian Center of Cardiology, P. Stradina University Hospital, Riga, Latvia
- University Malay Medical Center, Kuala Lumpur, Lembah Pantai, Malaysia
- Netherlands (4):
  - Het Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - AMC, Amsterdam
  - Amphia Hospital, Breda
  - St. Antonius Ziekenhuis, Nieuwegein
- Norway (2):
  - Haukeland university hospital, Bergen
  - Feiringklinikken AS, Feiring
- Poland (2):
  - Polsko Amerykanskie-Kliniki Serca American Heart, Ustroń
  - Institute of Cardiology, Warsaw
- Portugal (3):
  - Hospital Santa Maria, Lisbon
  - Hospitalar Santa Marta, Lisbon
  - Hospital São João, Porto
- Bakulev Scientific Center for Cardiovascular Surgery, Moscow, Russia
- South Africa (2):
  - Bloemfontein Medi-Clinic, Bloemfontein
  - Unitas Hospital, Pretoria
- Spain (5):
  - Hospital General de Alicante, Alicante
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clinico San Carlos, Hemodynamics Department, Madrid
  - H. Miguel Servet. Zaragoza, Cardiology Service, Zaragoza
- Switzerland (3):
  - Inselspital Bern, Kardiologie, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Cardiocentro Ticino, Lugano
- United Kingdom (4):
  - Queen Elizabeth Hospital, London
  - Freeman Hospital, London
  - Hammersmith Hospital, London
  - St Mary's Hospital, London
- Venezuela (2):
  - Centro Medico de Caracas, Caracas
  - Clinica Santa Sofia, Caracas

REFERENCES:
- [Background] Morice MC. XIENCE V SPIRIT WOMEN clinical trial: characterization of the female population undergoing stent implantation. Womens Health (Lond). 2008 Sep;4(5):439-43. doi: 10.2217/17455057.4.5.439. PMID 19072483
- [Derived] Genereux P, Rutledge DR, Palmerini T, Caixeta A, Kedhi E, Hermiller JB, Wang J, Krucoff MW, Jones-McMeans J, Sudhir K, Simonton CA, Serruys PW, Stone GW. Stent Thrombosis and Dual Antiplatelet Therapy Interruption With Everolimus-Eluting Stents: Insights From the Xience V Coronary Stent System Trials. Circ Cardiovasc Interv. 2015 May;8(5):e001362. doi: 10.1161/CIRCINTERVENTIONS.114.001362. PMID 25940520